CLINICAL TRIAL: NCT05586282
Title: Role of Candidate Proteins in Capillary Leakage During Acute Circulatory Failure
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APH211381
Record Dates: First submitted 2022-10-11; First posted 2022-10-19 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cardiogenic Shock; Postresuscitation Disease; Septic Shock
MeSH Terms: conditions — Shock, Cardiogenic; Post-Cardiac Arrest Syndrome; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples (serum and Ficoll-isolated cells), taken as part of the study will be stored in a biological sample collection (for patient who have given their consent).
  * ELISA dosage of candidate proteins and inflammation cytokines (IL-1, IL-6, TNF-alpha, IL-10, IL-33, angiopoïétine 2, E-sélectine) + further analysis (not described in the protocol) which may be useful in light of advances in scientific knowledge
  * For FACs and RNA sequencing + further analysis (not described in the protocol) which may be useful in light of advances in scientific knowledge
  * Immuno-inflammatory analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with a circulatory failure: All patients hospitalized in ICU with a circulatory failure due to septic shock, cardiogenic shock, or post-resuscitation syndrome.

SUMMARY:
* Testing the association between circulating candidate proteins and the level of vascular leakage for three distinct forms of circulatory failure: cardiogenic shock, septic shock, and post-resuscitation syndrome.
* Describing immuno-inflammatory profiles associated with massive vascular leakage during those three forms of circulatory failure in humans

DETAILED DESCRIPTION:
Circulatory shocks are responsible for one third of intensive care unit (ICU) admissions (20,000 patients per year in France) and are associated with 40% mortality [1,2]. Vascular hyperpermeability (also called vascular leakage) is a major feature of circulatory failure. During systemic inflammatory response syndrome (SIRS), massive vascular leakage affects macro and micro-circulation, and participates in the development of multiple organ failure [1,3]. Accordingly, fluid balance (the difference between fluid input and output) correlates independently with mortality during both septic and cardiogenic shock [4-7] and controlling capillary leakage was highly beneficial in numerous animal models of circulatory failure [8-10]. However, the determinants of vascular leakage remain poorly understood in humans.

The purpose of this study is to evaluate the link between circulatory levels of several proteins and the level of vascular leakage, in three distinct types of circulatory shocks.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent from patient or a legal representative/family member/close relative. The patient will be asked to give his/her consent for the continuation of the trial when his/her condition will allow.
2. Affiliation to social security (AME excluded)
3. Patient with one of the circulatory failures described below:

   * septic shock
   * cardiogenic shock
   * post-resuscitation syndrome
   * Cardiogenic shock:

     * Need for a catecholamine support to maintain mean arterial pressure>65 mmHg, AND
     * Cardiac index <2 L/min/m2 or left ventricular ejection fraction (LVEF)<35%, AND
     * Lactate >2.0 mmol/l
   * Post-resuscitation syndrome:

     * Cardiac arrest (absence of spontaneous respiration, palpable heartbeat, and responsiveness to stimuli> 1 min) with a compatible electrocardiogram (asystole/pulseless electrical activity/ventricular tachycardia), AND
     * Need for a catecholamine support to maintain mean arterial pressure>65 mmHg, AND
     * Lactate >2.0 mmol/l
   * Septic shock:

     * Suspected or proven bacterial infection
     * Need for a vasopressor support to maintain mean arterial pressure>65 mmHg
     * Lactate >2.0 mmol/l
     * Cardiac index>3L/min/m2 or LVEF>40%

Exclusion Criteria:

1. Onset of shock (catecholamine infusion) >12 hours prior to inclusion
2. Age <18 year old
3. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients hospitalized in ICU with a circulatory failure due to septic shock, cardiogenic shock, or post-resuscitation syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Fluid balance from Day 0 to day 3 | Between Day 0 and Day 3
  (ml/kg of initial body weight). The fluid balance, routinely monitored in ICU, represents fluid intakes (perfusion, oral intakes,..) - fluid losses (diuresis, diarrhea,…)

SECONDARY OUTCOMES:
Fluid balance | Day 1, Day 3, Day 7, Day 14
  (ml/kg of initial body weight). The fluid balance, routinely monitored in ICU, represents fluid intakes (perfusion, oral intakes,..) - fluid losses (diuresis, diarrhea,…)
Extra-vascular lung water index | Day 0, Day 1, Day 3, Day 7, Day 14
  Extra-vascular lung water index (EVLWi, ml/kg) and pulmonary vascular permeability index measured by transpulmonary thermodilution at corresponding time-points
Serum albuminemia | Day 0, Day 1, Day 3, Day 7, Day 14
  g/L
Serum lactatemia | Day 0, Day 1, Day 3, Day 7, Day 14
  mmoles/L
Arterial PaO2 | Day 0, Day 1, Day 3, Day 7, Day 14
  (mmHg)
Circulating cytokine inflammatory profile IL-33 | Day 0, Day 1, Day 3, Day 7, Day 14
  (pg/ml)
Circulating cytokine inflammatory profile TNF-alpha | Day 0, Day 1, Day 3, Day 7, Day 14
  (pg/ml)
Circulating cytokine inflammatory profile IL-6 | Day 0, Day 1, Day 3, Day 7, Day 14
  (pg/ml)
Circulating cytokine inflammatory profile IL-1 | Day 0, Day 1, Day 3, Day 7, Day 14
  (pg/ml)
SOFA score | Day 0, Day 1, Day 3, Day 7, Day 14
  Association between circulating candidate proteins, the immune-inflammatory profile of the patients and SOFA score
Catecholamine-free days | Day 0 to Day 7, Day 30
  Number of days alive without receiving any catecholamine
Ventilatory-free days | Day 0 to Day 7, Day 30
  Number of days alive without receiving any machenical ventilation, invasive or non-invasive
Renal replacement therapy-free | Day 0 to Day 7, Day 30
  Number of days alive without receiving any renal replacement therapy
Mortality | Day 30

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Européen Georges Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: No